CLINICAL TRIAL: NCT05868746
Title: Measuring Breast Cancer Survivor's Subjective Responses to Exercise Using a Novel, Smartwatch-based EMA Method: A Pilot Study
Brief Title: An Observational Pilot Study to Test a Smartwatch-based EMA Method During Exercise With Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Courtney J. Stevens, Assistant Professor of Psychiatry, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02000934_1B; IRG-21-136-36-IRG (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2023-05-09; First posted 2023-05-22 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this pilot study is to evaluate the feasibility and acceptability of collecting ecological momentary assessment data regarding feeling states during physical activity among a cohort of breast cancer survivors, using a novel smartwatch app created by the study team called "PHITbit."

ELIGIBILITY:
Inclusion Criteria:

* Within 5 years of completing primary cancer treatment (surgery, chemotherapy, and radiation) for Stage 0-III breast cancer.
* Own an Android or iPhone smartphone and willing to use the smartphone to complete app-based surveys during the assessment period.
* Willing to wear the ActiGraph monitor during the assessment period.
* Willing to wear the study issued Fitbit Versa 3 smartwatch during the assessment period.
* Access to internet to complete REDCap survey assessments.

Exclusion Criteria:

* Non-English speaking/not able to read English.
* Evidence of major contraindications for exercise per the 2020 Physical Activity Readiness-Questionnaire (PAR-Q)+.
* Currently pregnant.
* History of severe mental illness or currently taking mood stabilizing medications (antipsychotics, anticonvulsants, or lithium).
* Evidence of moderate-severe depressive symptoms (indicated by a score ≥ 10 on Patient Health Questionnaire-8). -Evidence of moderate-severe cognitive impairment (indicated by a score < 3 on a 6- item cognitive screener).
* Evidence of clinically significant substance use as indicated by a score of ≥ 2 on the CAGE-AID screener.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients under the care of a Dartmouth Cancer Center oncology provider.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of using a smartwatch-based ecological momentary assessment (EMA) method during exercise measured as the proportion of participants who use the data collection app and provided at least 3 responses to EMAs during a single exercise session. | 10 day data collection period
  The number of participants who use the smartwatch data collection app and respond to at least 3 EMAs during a single exercise session at least once during the 10-day data collection period out of the total number of participants enrolled at the end of the10-day data collection period.
Acceptability of collecting during-exercise feeling state data using a smartwatch-based ecological momentary assessment method measured using the System Usability Scale. | End of study follow-up (post 10-day data collection period)
  The System Usability Scale (SUS) is a 10-item self-report scale used to measure perceived usability of a system, method, or tool. Responses on the SUS range from 1 = strongly disagree to 5 = strongly agree. Higher scores indicate greater acceptability.
Acceptability of collecting during-exercise feeling state data using a smartwatch-based ecological momentary assessment method measured via a semi-structured interview. | End of study follow-up (post 10-day data collection period)
  Semi-structured interview to assess participants' perceptions regarding their experience using the smartwatch-based ecological momentary assessment method.

SECONDARY OUTCOMES:
Proportion of the sample with valid accelerometer data at the end of the 10-day data collection period. | 10 day data collection period
  The number of participants with valid accelerometer data out of the total number of participants in the sample during the 10-day data collection period.
Rate of phone-based ecological momentary assessment (EMA) prompt completion. | 10 day data collection period
  The number of phone-based EMA survey prompts completed by participants during the 10-day data collection period out of the total number of phone-based EMA survey prompts delivered to participants.
Rate of electronic daily dairy completion. | 10 day data collection period
  The number of electronic daily dairies completed by participants during the 10-day data collection period out of the total number of electronic daily dairies delivered to participants.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney J Stevens, PhD, Principal Investigator — Dartmouth-Hitchcock Health
Locations (1):
- Dartmouth-Hitchcock Clinic, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No